CLINICAL TRIAL: NCT04513548
Title: A Two-part Exploratory Study Combining a Pilot Study in Healthy Subjects and Chronic Spontaneous Urticaria Patients (Part 1) and a Randomized, Subject, Investigator and Sponsor-blinded, Placebo Controlled, Study (Part 2) to Assess the MechAniSm of acTion of ligElizumab (QGE031) in Patients With Chronic uRticaria (MASTER)
Brief Title: Study of Mechanism of Action of Ligelizumab (QGE031) in Patients With Chronic Urticaria
Acronym: MASTER
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CQGE031C2203; 2019-001048-24 (EudraCT Number)
Record Dates: First submitted 2020-08-07; First posted 2020-08-14 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Chronic Spontaneous Urticaria; Cholinergic Urticaria; Cold Urticaria
Keywords: chronic spontaneous urticaria; chronic inducible urticaria; cholinergic urticaria; cold urticaria; ligelizumab (QGE031)
MeSH Terms: conditions — Chronic Urticaria; Cold Urticaria; Chronic Inducible Urticaria | interventions — ligelizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Part 1 is not masked Part 2 is masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ligelizumab (Experimental): test drug
  Interventions: Drug: Ligelizumab
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ligelizumab — One injection every four weeks
  Arms: Ligelizumab
Drug: Placebo — One injection every four weeks
  Arms: Placebo

SUMMARY:
The purpose of the study is to investigate the mechanism of action for ligelizumab (QGE031) treatment in patients with chronic urticaria.

The study has two parts. The study population will consist of approximately 68 male and female healthy volunteers and patients. In Part 1, approximately 20 healthy volunteers and patients with chornic urticaria will be enrolled. In Part 2 approximately 48 patients with chronic urticaria (spontaneous chronic urticaria, cholinergic urticaria or cold urticaria). Part 1 consists of a screening period up 2 weeks and a visit with skin tests; there is no treatment taken in Part 1. Part 2 is randomized, subject, investigator and sponsor blinded. It consists of a screening period up to 4 weeks, a 16 week treatment period and a 12-week follow-up period after last treatment. A follow-up call at Week 32 will be performed via telephone.

DETAILED DESCRIPTION:
There are 58 patients out of 68 participants (10 are Healthy Volunteers)

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers • Healthy male and female subjects in good health as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at screening.

CSU and CINDU patients (cold and cholinergic urticaria)

• Part 2: Positive response to challenge test with ciprofloxacin 250 mg/ml or 125 mg/ml, defined as a wheal formation with longest diameter of at least 3 mm and middle perpendicular diameter of at least 2 mm at Day 1.

CSU patients

* Diagnosis of CSU, not adequately controlled with H1-AH at approved doses alone at the time of randomization, as defined by all of the following:
* UAS7 score (range 0-42) ≥ 16 and HSS7 (range 0-21) ≥ 8 during 7 days prior to randomization
* CSU for ≥ 6 months CINDU patients (cold and cholinergic urticaria)
* For patients with cold urticaria: Cold urticaria symptoms persisting for at least 6 months prior to study enrollment and a positive cold urticaria provocation test defined as wheal response to TempTest 4.0® at Day 1.
* For patients with cholinergic urticaria: Cholinergic urticaria symptoms for at least 6 months prior to enrollment and a positive response in the challenge test defined as a wheal response in the pulse controlled ergometry provocation test (30 minutes bicycle challenge) at Day 1

Exclusion Criteria:

Healthy volunteers

* History of allergies or allergy to the challenge substances including ciprofloxacin, icatibant, other quinolones or excipients of the substances being used in the study.
* Recent (within the last three years) and/or recurrent history of autonomic dysfunction (e.g. recurrent episodes of fainting, palpitations, etc.).
* Donation or loss of 450 mL or more blood within eight weeks prior to initial dosing, or longer if required by local regulations.

CSU and CINDU patients (cold and cholinergic urticaria)

* History of allergies or allergy to the challenge substances including ciprofloxacin, icatibant (Part 1 only), other quinolones or excipients of the substances being used in this study.
* Contraindications to or hypersensitivity to antihistamines (such as fexofenadine, loratadine, cetirizine, rupatadine, bilastine) or epinephrine or any of the ingredients.
* History or presence of renal disease and/or estimated glomerular filtration (eGFR) rate of < 35 mL/min as calculated by the CKD-EPI formula at Screening.
* For subjects who enter Part 2: Patients with a history of or a risk of parasite infections (recent stay in tropical/subtropical areas with low hygiene standards). To allow enrollment of a patient at risk perform stool examinations for ova or parasites and demonstrate absence of infection first.
* Diseases with possible signs and symptoms of urticaria or angioedema such as urticarial vasculitis, erythema multiforme, cutaneous mastocytosis (urticaria pigmentosa), and hereditary or acquired angioedema (e.g. due to C1 inhibitor deficiency).

CSU patients • Clearly defined underlying etiology for chronic urticaria symptoms other than CSU. This includes the following: CSU patients should not have inducible urticaria forms impacting their daily symptoms in a relevant way, such as but not limited to urticaria factitia, cold-, heat-, solar-, pressure-, delayed pressure, aquagenic-, cholinergic-, or contact-urticaria.

CINDU patients (cold and cholinergic urticaria)

• Clearly defined underlying etiology for chronic urticaria symptoms other than CINDU. This includes the following: CINDU patients should not have spontaneous urticaria impacting their symptoms in a relevant way.

Other protocol-defined inclusion/exclusion criteria may apply .

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2022-07-19 (Actual)

PRIMARY OUTCOMES:
Part 1: Wheal and erythema size after skin prick test with several different ciprofloxacin and icatibant concentrations. | At Day 1
  Size of the wheal and erythema in mm will be measured after the skin prick and intradermal tests are performed. Different dilution steps will be applied (to differentiate Chronic Spontaneous Urticaria patients and healthy controls) for ciprofloxacin and icatibant to determine the conditions to be used in Part 2.
Part 2: Change in wheal size after challenge procedure from Day 1 (pre-dose) to week 16. | Day 1 and Week 16
  Size of wheal in mm2 after skin prick test and autologous serum skin test will be measured.

SECONDARY OUTCOMES:
Part 2: Urticaria Control Test | Day 1, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28
  The Urticaria Control Test (UCT) is a questionnaire that assesses the extent of the disease control over the previous 4 weeks. It consists of 4 questions, each rated from 0 to 4 points. Subsequently, the scores for all 4 questions are summed up. The minimum and maximum UCT scores are 0 and 16, with 12 points or higher indicating controlled disease, and 16 points indicating complete disease control.
Part 2: Weekly Urticaria Activity Score | Throughout the study (to 28 weeks)
  Chronic Spontaneous Urticaria (CSU) patients: The Urticaria Activity Score (UAS) is evaluated in the screening period and throughout the study. It records each morning and evening on a daily basis symptoms of itch and hives into a patient diary. The UAS is a composite score with numeric severity intensity ratings on a scale of 0 - 3 for the number of wheals (hives) and the itch intensity. The UAS7 is the sum of the daily UAS scores over 7 days. UAS7 values range from 0 to 42, with higher values indicate higher disease activity.
Part 2: Cholinergic Urticaria Activity score | Day 1 to Week 28
  Cholinergic urticaria patients: Cholinergic Urticaria Activity score (CholUAS) is a questionnaire that records each evening on a daily basis symptoms of itch and hives and the general assessment of disease severity into a patient diary. The CholUAS is a composite score with numeric ratings on a scale of 0 - 3 for the intensity of wheals (hives), the itch intensity, and the overall assessment of the disease severity. The total score is a sum of scores multiplied with the score for the trigger. The CholUAS7 is the sum of the daily CholUAS scores over 7 days. Higher values indicate a higher disease activity.
Part 2: Chronic Urticaria Quality of Life questionnaire | Day 1, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28
  CSU patients: The Chronic Urticaria Quality of Life questionnaire (CU-Q2oL) is a questionnaire that measures the relative burden of chronic urticaria on subjective well-being. It consists of 23 questions in 3 domains (symptoms, general impairment, difficulties and problems due to urticaria). with a total score of 0 to 100 %. Higher scores indicate higher impairment in quality of life.
Part 2: Angioedema control test | Day 1, Week 16, Week 28
  CSU patients with angioedema: Angioedema Control Test (AECT) is a questionnaire that assesses the extent of the symptom control (angioedema). It consists of 4 questions, each rated from 0 to 4 points. Subsequently, the scores for all 4 questions are summed up. The minimum and maximum AECT scores are 0 and 16, with 10 points or higher indicating controlled disease, and 16 points indicating complete disease control.
Part 2: Cholinergic Urticaria Quality of Life questionnaire | Day 1, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28
  Cholinergic patients: The Cholinergic Urticaria Quality of Life questionnaire (Chol-Q2oL) is a questionnaire that measures the relative burden of cholinergic urticaria on subjective well-being. The questionnaire consists of 28 items, each item being scored between 0 and 4. Higher scores indicate higher impairment in quality of life.
Part 2: Provocation test for cholinergic patients | Day 1, Week 4, Week 16, Week 28
  Cholinergic patients: Time from onset of sweating and urticaria symptoms after an exercise on a stationary bicycle.
Part 2: Temperature trigger test for cold urticaria patients | Day 1, Week 4, Week 16, Week 28
  Cold urticaria patients: The temperature that will provoke the formation of wheals will be assessed.
Part 2: Number of patients with adverse events | Throughout the study (to 28 weeks)
  Part 2: Safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: Results for CQGE031C2203 from the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18055
- See also: Patient Lay Trial Summary — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1543